CLINICAL TRIAL: NCT02931838
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Phase 2 Study to Evaluate the Clinical Efficacy and Safety of BMS-986165 in Subjects With Moderate to Severe Psoriasis
Brief Title: Study to Evaluate Effectiveness and Safety in Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-011
Record Dates: First submitted 2016-10-03; First posted 2016-10-13 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BMS-986165 Dose 1 (Experimental): Specified dose of BMS-986165 on specified days.
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 2 (Experimental): Specified dose of BMS-986165 on specified days.
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 3 (Experimental): Specified dose of BMS-986165 on specified days.
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 4 (Experimental): Specified dose of BMS-986165 on specified days.
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 5 (Experimental): Specified dose of BMS-986165 on specified days.
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator): Specified dose of Placebo for BMS-986165 on specified days.
  Interventions: Drug: Placebo for BMS-986165

INTERVENTIONS:
Drug: BMS-986165
  Arms: BMS-986165 Dose 1; BMS-986165 Dose 2; BMS-986165 Dose 3; BMS-986165 Dose 4; BMS-986165 Dose 5
Drug: Placebo for BMS-986165
  Arms: Placebo

SUMMARY:
A Study to evaluate efficacy and safety in subjects with moderate to severe Psoriasis treated with BMS-986165

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male and female, ages 18 to 70 years
* Diagnosis of plaque psoriasis for 6 months
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test, must not be pregnant, lactating, breastfeeding or planning pregnancy
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of the study drug plus 90 days.

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate oral medication
* Positive hepatitis-B (HBV) surface antigen
* Positive hepatitis-C (HCV) antibody
* Any history or risk for tuberculosis (TB)
* Any major illness/condition or evidence of an unstable clinical condition
* Chest X-ray findings suspicious of infection at screening
* has received ustekinumab, secukinumab or ixekizumab within 6 months of first administration of study medication
* Has received anti-Tumor Necrosis Factor (TNF) inhibitor(s) within 2 months of first administration of study medication
* Has received Rituximab within 6 months of first administration of study medication
* Topical medications/treatments for psoriasis within 2 weeks of the first administration of any study medication
* Any systemic medications/treatments for psoriasis within 4 weeks of the first administration of any study medication

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (67):
- United States (16):
  - University of California Irvine, Irvine, California
  - University of California San Diego, San Diego, California
  - Renstar Medical Research, Ocala, Florida
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - PMG Research of Christie Clinic, LLC, Champaign, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dartmouth-Hitchcock Medical Center-Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Piedmont Plastic Surgery & Dermatology - Charlotte/Blakeney Location, Charlotte, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, PLC, Wilmington, North Carolina
  - Central Sooner Research, Norman, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Rivergate Dermatology Clinical Research Center, Pllc, Goodlettsville, Tennessee
  - Local Institution, Knoxville, Tennessee
  - Austin Dermatology Associates, Austin, Texas
- Australia (4):
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Wolloongabba, Queensland
  - Local Institution, Melbourne, Victoria
  - Local Institution, Nedlands, Western Australia
- Canada (11):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Markham, Ontario
  - Local Institution, Mississauga, Ontario
  - Local Institution, Peterborough, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Montreal, Quebec
- Germany (9):
  - Local Institution, Dresden
  - Local Institution, Gera
  - Local Institution, Hamburg
  - Local Institution, Kiel
  - Local Institution, Lübeck
  - Local Institution, Mahlow
  - Local Institution, Mainz
  - Local Institution, Schwerin
  - Local Institution, Stuttgart
- Japan (13):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Kamigyō-ku, Kyoto
  - Local Institution, Shimotsuke-shi, Tochigi
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Shinagawa-Ku, Tokyo
  - Local Institution, Shinjuku-ku, Tokyo
  - Local Institution, Skinjuku-ku, Tokyo
  - Local Institution, Kumamoto
  - Local Institution, Osaka
  - Local Institution, Tokyo
- Latvia (3):
  - Local Institution, Daugavpils
  - Local Institution, Riga
  - Local Institution, Ventspils
- Mexico (2):
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
- Poland (9):
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Osielsko
  - Local Institution, Siedlce
  - Local Institution, Skierniewice
  - Local Institution, Warsaw
  - Local Institution, Wroc?aw
  - Local Institution, Wroclaw

REFERENCES:
- [Derived] Catlett IM, Gao L, Hu Y, Banerjee S, Krueger JG. Pharmacodynamic Response to Deucravacitinib, an Oral, Selective, Allosteric TYK2 Inhibitor, in a Global, Phase 2, Randomized, Double-Blind, Placebo-Controlled Psoriasis Trial. Dermatol Ther (Heidelb). 2024 Oct;14(10):2827-2839. doi: 10.1007/s13555-024-01262-5. Epub 2024 Sep 16. PMID 39283417
- [Derived] Thaci D, Strober B, Gordon KB, Foley P, Gooderham M, Morita A, Papp KA, Puig L, Menter MA, Colombo MJ, Elbez Y, Kisa RM, Ye J, Napoli AA, Wei L, Banerjee S, Merola JF, Gottlieb AB. Deucravacitinib in Moderate to Severe Psoriasis: Clinical and Quality-of-Life Outcomes in a Phase 2 Trial. Dermatol Ther (Heidelb). 2022 Feb;12(2):495-510. doi: 10.1007/s13555-021-00649-y. Epub 2022 Jan 13. PMID 35025062
- [Derived] Catlett IM, Hu Y, Gao L, Banerjee S, Gordon K, Krueger JG. Molecular and clinical effects of selective tyrosine kinase 2 inhibition with deucravacitinib in psoriasis. J Allergy Clin Immunol. 2022 Jun;149(6):2010-2020.e8. doi: 10.1016/j.jaci.2021.11.001. Epub 2021 Nov 10. PMID 34767869
- [Derived] Papp K, Gordon K, Thaci D, Morita A, Gooderham M, Foley P, Girgis IG, Kundu S, Banerjee S. Phase 2 Trial of Selective Tyrosine Kinase 2 Inhibition in Psoriasis. N Engl J Med. 2018 Oct 4;379(14):1313-1321. doi: 10.1056/NEJMoa1806382. Epub 2018 Sep 11. PMID 30205746
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 268 participants were randomized in the study; One participant was randomized but did not receive study drug due to being lost to follow-up
Groups:
- Placebo: Placebo for BMS-986165
- BMS-986165 3MG QOD: BMS-986165 3mg capsules Every Other Day
- BMS-986165 3MG QD: BMS-986165 3mg capsules Every Day
- BMS-986165 3MG BID: BMS-986165 3mg capsules Twice Daily
- BMS-986165 6MG BID: BMS-986165 6mg capsules Twice Daily
- BMS-986165 12MG QD: BMS-986165 12mg capsules Every Day
Period: Overall Study
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Started | 45 | 44 | 44 | 45 | 45 | 44
Completed | 31 | 34 | 36 | 42 | 39 | 42
Not Completed | 14 | 10 | 8 | 3 | 6 | 2
Not completed — Reason not provided by investigator | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Poor/non-compliance | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 4 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 2 | 0
Not completed — Subject request to discontinue treatment | 4 | 3 | 3 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 2 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- BMS-986165 3MG QD: BMS-986165 3 mg capsules every day
- BMS-986165 3MG BID: BMS-986165 3 mg capsules twice daily
- BMS-986165 6MG BID: BMS-986165 6 mg capsules twice daily
- BMS-986165 12MG QD: BMS-986165 12 mg capsules every day
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD | Total
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized and treated participants
  Years | 46.4 (11.93) | 41.0 (11.8) | 45.0 (13.77) | 45.6 (15.10) | 42.8 (12.90) | 46.6 (11.62) | 44.6 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    Female | 8 | 8 | 14 | 19 | 10 | 14 | 73
    Male | 37 | 36 | 30 | 26 | 35 | 30 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized and treated participants
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 1 | 3
    Asian | 5 | 6 | 5 | 5 | 9 | 6 | 36
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 2
    White | 40 | 35 | 39 | 39 | 35 | 37 | 225
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Moderate to Severe Psoriasis Experiencing a 75% Improvement (Reduction From Baseline) in PASI Score (PASI-75 Response Rate) on Day 85 (Week 12)
Description: Psoriasis Area and Severity Index (PASI) 75 response: patients who achieved ≥ 75% improvement (reduction) in PASI score compared to baseline were defined as PASI 75 responders. PASI scores can range from 0, corresponding to no signs of psoriasis up to theoretical maximum of 72.0, which means a higher PASI score reflects a higher psoriasis activity.
Time Frame: Day 1 to Day 85
Population: All Randomized and Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Percentage | 6.7 [1.4 to 18.3] | 9.1 [2.5 to 21.7] | 38.6 [24.4 to 54.5] | 68.9 [53.4 to 81.8] | 66.7 [51.0 to 80.0] | 75.0 [59.7 to 86.8]
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3MG QOD; Test type: Superiority; p = 0.4873, Chi-squared — Nominal p-value; P-value is from the Fishers Exact if at least one cell count is <5. Otherwise, p-value is from the Chi-Square test
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 3MG QD; Test type: Superiority; p = 0.0003, Chi-squared — Nominal p-value; P-value is from the Fishers Exact if at least one cell count is <5. Otherwise, p-value is from the Chi-Square test
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 3MG BID; Test type: Superiority; p < 0.0001, Chi-squared — Nominal p-value; P-value is from the Fishers Exact if at least one cell count is <5. Otherwise, p-value is from the Chi-Square test
Statistical Analysis 4: Comparison: Placebo vs BMS-986165 6MG BID; Test type: Superiority; p < 0.0001, Chi-squared — Nominal p-value; P-value is from the Fishers Exact if at least one cell count is <5. Otherwise, p-value is from the Chi-Square test
Statistical Analysis 5: Comparison: Placebo vs BMS-986165 12MG QD; Test type: Superiority; p < 0.0001, Chi-squared — Nominal p-value; P-value is from the Fishers Exact if at least one cell count is <5. Otherwise, p-value is from the Chi-Square test

2. Secondary Outcome: Percentage of Participants on Day 85 With PASI-50, PASI-90, PASI-100.
Description: Percentage of patients achieving Psoriasis Area and Severity Index (PASI) 50, PASI 90 and PASI 100 responses on Day 85. PASI 50 response: patients who achieved ≥ 50% improvement (reduction) in PASI score compared to baseline were defined as PASI 50 responders. PASI 90 response: patients who achieved ≥ 90% improvement (reduction) in PASI score compared to baseline were defined as PASI 90 responders. PASI 100 response: patients who achieved ≥ 100% improvement (reduction) in PASI score compared to baseline were defined as PASI 100 responders. PASI scores can range from 0, corresponding to no signs of psoriasis up to theoretical maximum of 72.0, which means a higher PASI score reflects a higher psoriasis activity.
Time Frame: Day 1 to Day 85
Population: All Randomized and Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Percentage
  % of participants with PASI-50 at Day 85 | 31.1 [18.2 to 46.6] | 43.2 [28.3 to 59.0] | 68.2 [52.4 to 81.4] | 91.1 [78.8 to 97.5] | 77.8 [62.9 to 88.8] | 88.6 [75.4 to 96.2]
  % of participants with PASI-90 at Day 85 | 2.2 [0.1 to 11.8] | 6.8 [1.4 to 18.7] | 15.9 [6.6 to 30.1] | 44.4 [29.6 to 60.0] | 44.4 [29.6 to 60.0] | 43.2 [28.3 to 59.0]
  % of participants with PASI-100 at Day 85 | 0 [0.0 to 7.9] | 2.3 [0.1 to 12.0] | 0 [0.0 to 8.0] | 8.9 [2.5 to 21.2] | 17.8 [8.0 to 32.1] | 25.0 [13.2 to 40.3]

3. Secondary Outcome: Percentage of Participants on Day 85 With sPGA Score of 0 or 1 (sPGA0/1 Response Rate).
Description: Percentage of participants achieving a clear (0) or almost clear (1) status on the Static Physician Global Assessment (sPGA) on Day 85. This index evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The assessment was scored on a scale of 0 to 5, where 0 = clear, with no evidence of plaque elevation, erythema, or scale, and 5 = severe induration, erythema, and scaling.
Time Frame: Day 1 to Day 85
Population: All Randomized and Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Percentage | 6.7 [1.4 to 18.3] | 20.5 [9.8 to 35.3] | 38.6 [24.4 to 54.5] | 75.6 [60.5 to 87.1] | 64.4 [48.8 to 78.1] | 75.0 [59.7 to 86.8]

4. Secondary Outcome: Change From Baseline in DLQI Scores on Day 85
Description: The DLQI is a participant reported quality of life index which consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week. Each question is scored on a scale of 0 to 3 by a tick box: "not at all", "a little", "a lot", or "very much". The scores are summed, giving a range from 0 (no impairment of life quality) to 30 (maximum impairment)
Time Frame: Day 1 to Day 85
Population: All Randomized and Treated Participants
Measure: Mean (95% Confidence Interval); unit: Score
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Score | -2.85 [-4.33 to -1.37] | -3.76 [-5.15 to -2.38] | -6.07 [-8.07 to -4.08] | -9.67 [-11.42 to -7.93] | -8.38 [-10.72 to -6.03] | -10.16 [-12.27 to -8.06]

5. Secondary Outcome: Change From Baseline in BSA on Day 85
Description: Measurement of psoriasis body surface area (BSA) involvement is estimated using the handprint method with the size of a patient's handprint representing ~1% of body surface area involved.The total BSA = 100% with breakdown by body region as follows: head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), trunk including axillae and groin = 30% (30 handprints), lower extremities including buttocks = 40% (40 handprints). A decrease from Baseline indicates improvement. Change from Baseline was calculated as Baseline score - Day 85 score; a positive change from Baseline therefore indicates improvement.
Time Frame: Day 1 to Day 85
Population: All Randomized and Treated Participants
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Percentage | -7.71 [-11.88 to -3.54] | -5.50 [-8.17 to -2.83] | -12.59 [-18.28 to -6.89] | -18.60 [-23.69 to -13.52] | -17.23 [-20.85 to -13.60] | -15.16 [-18.64 to -11.69]

6. Secondary Outcome: Trough Observed Plasma Concentration of BMS-986165 (Ctrough)
Description: Pharmacokinetics of BMS-986165 were derived from plasma concentration versus time data. Ctrough= Trough observed plasma concentration
Time Frame: Days 8, 15, 29, 57, 85
Population: All participants who received any study medication and have any available concentration-time data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 44 | 44 | 44 | 45 | 44
ng/mL | 2.024 (3.7061) | 3.145 (3.1588) | 14.819 (9.1410) | 26.257 (14.6483) | 17.824 (22.7536)

7. Primary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of BMS-986195 as assessed by the number of subjects with adverse events (AEs); number of subjects with serious adverse events (SAEs); number of subjects with adverse events leading to discontinuation
Time Frame: Day 1 to day 115
Population: All Randomized and Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3MG QOD | BMS-986165 3MG QD | BMS-986165 3MG BID | BMS-986165 6MG BID | BMS-986165 12MG QD
Number analyzed (Participants) | 45 | 44 | 44 | 45 | 45 | 44
Participants
  No. of participants with SAEs | 1 | 1 | 1 | 1 | 0 | 0
  No. of participants with AEs | 24 | 26 | 25 | 29 | 36 | 34
  No. of participants discontinued due to AEs | 2 | 1 | 2 | 1 | 3 | 1

ADVERSE EVENTS:
Time Frame: 20 weeks (assessed up to November 16, 2017)
Description: All Serious Adverse Events were collected from the date of participant's written consent until 30 days post discontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. The collection of non-serious Adverse Event information began at initiation of study drug.Treatment Emergent AEs are determined from first dose to within 30 days after last dose.
Arm/Group | Placebo | BMS-986165 3mg QOD | BMS-986165 3mg QD | BMS-986165 3mg BID | BMS-986165 6mg BID | BMS-986165 12mg QD
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44 | 0/44 | 0/45 | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/44 | 1/44 | 1/45 | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 13/45 | 14/44 | 18/44 | 15/45 | 25/45 | 19/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | BMS-986165 3mg QOD (N=44) | BMS-986165 3mg QD (N=44) | BMS-986165 3mg BID (N=45) | BMS-986165 6mg BID (N=45) | BMS-986165 12mg QD (N=44)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | BMS-986165 3mg QOD (N=44) | BMS-986165 3mg QD (N=44) | BMS-986165 3mg BID (N=45) | BMS-986165 6mg BID (N=45) | BMS-986165 12mg QD (N=44)
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 4 | 0 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 5 | 5 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 1 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0 | 4 | 7
Blood immunoglobulin e increased (Investigations) | 1 | 3 | 2 | 0 | 2 | 3
Headache (Nervous system disorders) | 2 | 4 | 4 | 3 | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 3 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The limitations of this phase 2 trial include its small sample size and short duration; these results warrant confirmation in a larger trial of longer duration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02931838/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02931838/SAP_001.pdf